CLINICAL TRIAL: NCT04593732
Title: Clinical Investigation to Evaluate the STERN FIX Device As a Sternal Fixation System in Medium Sternotomy
Brief Title: STERN FIX Device As a Sternal Fixation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NEOS Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO-SC1-2020-01
Record Dates: First submitted 2020-10-05; First posted 2020-10-20 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Sternotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- STERN FIX (Sternal Stabilization System) (Experimental): Sternotomy closure with STERN FIX and supplemented with wires
  Interventions: Device: STERN FIX (Sternal Stabilization System)

INTERVENTIONS:
Device: STERN FIX (Sternal Stabilization System) — Sternotomy closure with STERN FIX and supplemented with wires

SUMMARY:
Pre-market clinical research, prospective, single-arm that aims to assess the sternal sealing in patients in which the sternum has been fixed with the STERN FIX system.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old.
* Patient who must have surgery in which a medium sternotomy is indicated.
* Subjects able to give their voluntary informed consent to participate in clinical research and from which written consent has been obtained.
* The subject is able to meet the requirements of the protocol and is willing to do so.

Exclusion Criteria:

* Patient with suspicious or known allergies or intolerance to implant material (PEEK - polyetheretherketone).
* Patient with limitations in blood supply, insufficient bone quantity or quality, severe osteoporosis, osteomalacia or other serious bone structural damage, which, at the surgeon's discretion, may interfere with the implantation or proper functioning of the product.
* Degenerative bone diseases.
* Patients with a latent or active infection or inflammation in the operating area that, at the surgeon's discretion, may interfere with the implantation or proper functioning of the product.
* Patients with fever or leukocytosis.
* Patient with spinal abnormalities that, according to the surgeon's discretion, prevent the use of the product, such as bone tumors located in the implant region.
* Patients who are pregnant or interested in becoming pregnant within 6 months of surgery.
* Nursing patients.
* Patients with life expectancy less than 6 months.
* Patients who are participating in or participating in the previous 4 weeks in another interventional clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Sternal stability according to clinical evaluation | 1 month post-surgery
  sternal instability scale (SIS) grade: from 0 (Clinically stable sternum ) to 3 Completely separated sternum

SECONDARY OUTCOMES:
sternal stability according to clinical evaluation | 7 days post-surgery, 6 months
  sternal instability scale (SIS) grade: from 0 (Clinically stable sternum ) to 3 Completely separated sternum
Prevalence of patients with dehiscence (without infection) | 6 months
Prevalence and causality of adverse events | 6 months
Prevalence of device deficiencies | 6 months
Prevalence of reinterventions | 6 months
Prevalence of superficial and deep sternal wound infections | 6 months
Prevalence of patients with compromised sternal integrity | 6 months
Prevalence of artefacts associated with the product in medical images | 6 months
Time to close the sternal (minutes) | surgery
Surgeon satisfaction score | immediately post-surgery
  Likert scale [1-5]
Chest Pain | pre-surgery, 7 days post-surgery, 1 month, 6 months
  Numeric Rating Scale [0-10]
Upper limb functionality | pre-surgery, 7 days post-surgery, 1 month, 6 months
  Upper Limb Functional Index (spanish version) score (0-100%)
Quality of life measured with EuroQol-5D-5L | pre-surgery, 7 days post-surgery, 1 month, 6 months
  EuroQol-5D-5L
Working status | pre-surgery, 6 months
  [Fully employed/ Working with restrictions/ Unemployed/ On sick leave/ Retired]
Sternal healing grade according to CT results | 6 months
  Healing score, between 0: No sign of healing, nonunion and 5: complete synthesis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No